CLINICAL TRIAL: NCT06443463
Title: A Phase 2, Global, Multicenter, Long-term Safety Study Designed to Assess the Safety and Tolerability of BHV-7000 in Subjects With Refractory Focal Onset Epilepsy
Brief Title: Long-term Safety and Tolerability of BHV-7000
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BHV7000-201; 2023-508813-18-00 (EU CTIS Number)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Focal Epilepsy
Keywords: Focal Epilepsy; Epilepsy; Seizure; Refractory Epilepsy; Partial Epilepsy
MeSH Terms: conditions — Epilepsies, Partial; Epilepsy; Seizures; Drug Resistant Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-7000 50 mg (Experimental)
  Interventions: Drug: BHV-7000
- BHV-7000 75 mg (Experimental)
  Interventions: Drug: BHV-7000

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 50 mg. Participants will take open-label investigational product (IP) once daily
  Arms: BHV-7000 50 mg
Drug: BHV-7000 — BHV-7000 75 mg. Participants will take open-label investigational product (IP) once daily
  Arms: BHV-7000 75 mg

SUMMARY:
A study to determine if BHV- 7000 is safe and tolerable in adults with refractory focal onset epilepsy

ELIGIBILITY:
Key Inclusion Criteria:

* Subjects who completed the double-blind phase (DBP) of prior parent study, BHV7000-302 or BHV7000-303.
* (FOCBP) Females of Child Bearing Potential must have a negative urine pregnancy test at the Baseline/Day 0 visit

Key Exclusion Criteria:

* Any condition, such as an ongoing AE with/without sequelae, or is poorly tolerating IP in the double-blind phase of the parent study, that would interfere with the subject's ability to comply with study instructions, place the subject at unacceptable risk, and/or confound the interpretation of safety or efficacy data from the study, as judged by the Investigator.
* Any medical condition, based on the judgement of the Investigator, that would confound the ability to adequately assess safety and efficacy outcome measures

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2024-07-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Deaths, Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and moderate or severe AEs | Up to 104 weeks
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with deaths, SAEs, AEs leading to discontinuation, and moderate and severe AEs.
Number of Subjects with Clinically Significant Laboratory Abnormalities | Up to 104 weeks
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 or 4 laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (281):
- United States (115):
  - Accel Research, Birmingham, Alabama
  - Onyx Clinical Trials, Peoria, Arizona
  - Xenoscience, Inc., Phoenix, Arizona
  - University of Arizona / Banner University Medical Center Phoenix, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - ARENSIA Exploratory Medicine, Phoenix, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - WRN, Rogers, Arkansas
  - University of California San Diego, La Jolla, California
  - Amicis Research Center, Lancaster, California
  - Memorialcare Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - University of California, Los Angeles, Los Angeles, California
  - Tri Valley Neurology Medical Associates, Inc., Mission Hills, California
  - Stanford University, Palo Alto, California
  - Profound Research LLC, Pasadena, California
  - Profound Research LLC, Poway, California
  - Kaiser Permanente, Aurora, Colorado
  - University of Colorado Anschultz Medical Campus, Aurora, Colorado
  - UConn Health, Farmington, Connecticut
  - Yale School of Medicine - Yale-New Haven Hospital, New Haven, Connecticut
  - EZR Research LLC, Boca Raton, Florida
  - Nova Clinical Research, LLC, Bradenton, Florida
  - Las Mercedes Medical Research, Hialeah, Florida
  - Coral Clinic Research, Homestead, Florida
  - University of Florida (Jacksonville), Jacksonville, Florida
  - Dm Healthworks, Kissimmee, Florida
  - University of Miami, Miami, Florida
  - Y&L Advance Health Care, Inc d/b/a Elite Clinical Research, Miami, Florida
  - Serenity Research Center, Miami, Florida
  - Floridian Research Institute, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Research Institute of Orlando, Orlando, Florida
  - Comprehensive Neurology Clinic, Orlando, Florida
  - Panhandle Research & Medical Clinic, Pensacola, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Knight Neurology, Rockledge, Florida
  - PENS, Tampa, Florida
  - Santos Research Center, Tampa, Florida
  - Encore Medical Research of Weston LLC., Weston, Florida
  - Pediatrix Medical Group of Florida, Winter Park, Florida
  - Augusta University, Augusta, Georgia
  - Accelerated Clinical Trials, LLC, Peachtree Corners, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Consultants in Epilepsy & Neurology, PLLC, Boise, Idaho
  - Northwestern University, Chicago, Illinois
  - Revive Research Institute, Inc., Elgin, Illinois
  - McFarland Clinic, Ames, Iowa
  - Bluegrass Epilepsy Research, Lexington, Kentucky
  - OLOLRMC, Baton Rouge, Louisiana
  - DelRicht Research, Baton Rouge, Louisiana
  - Neurocare Of Louisiana, Covington, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - LSU Health Shreveport, Shreveport, Louisiana
  - John Hopkins University, Baltimore, Maryland
  - Mid-Atlantic Epilepsy & Sleep Center, LLC, Bethesda, Maryland
  - Javara, Silver Spring, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Boston Neuro Research, South Dartmouth, Massachusetts
  - SRI International, Plymouth, Michigan
  - Revive Research Institute, Inc., Rochester Hills, Michigan
  - Minnesota Epilepsy Group, P.A., Roseville, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Somnos Clinical Research, Lincoln, Nebraska
  - NEREG, Hackensack, New Jersey
  - Inst of Neurology, Livingston, New Jersey
  - Tekton Research, Marlboro, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Dent Neurosciences Research Center, Amherst, New York
  - Northwell Health, Great Neck, New York
  - BCHP, Hawthorne, New York
  - Northwell Health, New Hyde Park, New York
  - NYU Langone Health, New York, New York
  - NYU, New York, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Montefiore Medical Center, The Bronx, New York
  - Five Towns Neuroscience Research, Woodmere, New York
  - UNC-Chapel Hill, Chapel Hill, North Carolina
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Accellacare, Mooresville, North Carolina
  - Wake Forest Baptist, Winston-Salem, North Carolina
  - NeuroScience Research Center, Canton, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - OSU, Columbus, Ohio
  - Wright State University, Dayton, Ohio
  - Oregon Neurology Associates, Springfield, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - AHN, Pittsburgh, Pennsylvania
  - UPMC, Pittsburgh, Pennsylvania
  - MUSC, Charleston, South Carolina
  - WR-ClinSearch, Chattanooga, Tennessee
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Horizon Clinical Research Group, Cypress, Texas
  - Clinical Research Solutions LLC, Cypress, Texas
  - Neurology Consultants of Dallas, PA, Dallas, Texas
  - M3 Wake Research-Dallas, Dallas, Texas
  - ANESC Research, El Paso, Texas
  - Tarrant Neurology Consultants, Fort Worth, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - UTHealth Houston, Houston, Texas
  - UTHSC, Houston, Texas
  - Stryde Research, Plano, Texas
  - UT Health San Antonio, San Antonio, Texas
  - Road Runner Research, Ltd, San Antonio, Texas
  - Intermountain Health, Murray, Utah
  - University of Utah, Salt Lake City, Utah
  - UVM MC, Burlington, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Medstar Health Research Institute, McLean, Virginia
  - Henrico Doctors Neurology Associates, LLC, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
- Argentina (10):
  - STAT Research S.A., Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital General de Agudos Dr. José María Ramos Mejia, Balvanera, Ciudad Autónoma de BuenosAires
  - Centro de Educación Médica e Investigaciones Clínicas Norberto Quirno CEMIC-Elías Galván 4102, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Hospital Británico de Buenos Aires, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Investigaciones Sanatorio Del Sur, San Miguel de Tucumán, Tucumán Province
  - Sanatorio de la Trinidad - Mitre, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Fundación Para La Lucha Contra Las Enfermedades Neurológicas de La Infancia - FLENI, Buenos Aires
  - Instituto Privado Kremer, Córdoba
  - Conci Carpinella - Santa Rosa N° 748, Córdoba
- Australia (8):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Brisbane & Women's Hospital, Herston, Queensland
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
  - Austin Health, Heidelberg, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Flinders Medical Centre, Bedford Park
- Austria (4):
  - Kepler Universitätsklinikum Linz - Med Campus III, Linz, Upper Austria
  - Christian Doppler-Klinik - Universitätsklinikum der PMU, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
- Belgium (5):
  - UZ Antwerpen, Edegem, Antwerpen
  - Hôpital Erasme, Anderlecht, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
  - CHU UCL Namur - Site Godinne, Yvoir, Namur
  - UZ Gent, Ghent, Oost-Vlaanderen
- Chile (5):
  - Centro de especialidades médicas Vanguardia, Temuco, Región de la Araucanía
  - Instituto Neurologico Thalamus, Viña del Mar, Región de Valparaíso
  - Hospital Padre Hurtado, Santiago, Región-MetropolitanadeSantiago
  - BIOCINETIC Ltda, Santiago, Región-MetropolitanadeSantiago
  - Centro de Investigacion Clinica UC, Santiago, Región-MetropolitanadeSantiago
- Croatia (5):
  - Clinical Hospital Dubrava, Zagreb, City of Zagreb
  - Clinical Hospital Sveti duh, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Sestre Milosrdnice - Vinogradska cesta 29, Zagreb, City of Zagreb
  - Klinicki bolnicki centar Zagreb, Zagreb, City of Zagreb
  - Clinical Hospital Center Rijeka - PPDS, Rijeka
- Czechia (2):
  - Fakultni nemocnice v Motole, Prague, Praha, Hlavní Mesto
  - Fakultni nemocnice u sv. Anny v Brne, Brno, South Moravian
- Denmark (3):
  - Odense Universitetshospital, Odense, Fyn
  - Aarhus University Hospital, Aarhus
  - Epilepsihospitalet Filadelfia, Dianalund
- Finland (3):
  - Kuopion yliopistollinen sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Helsinki University Hospital, Helsinki, Uusimaa
- France (9):
  - CHU de Strasbourg - Hôpital de Hautepierre, Strasbourg, Bas-Rhin
  - CHU Dijon Bourgogne, Dijon, Côte-d'Or
  - CHU de Toulouse-Hôpital Pierre-Paul Riquet-Site de Purpan, Toulouse, Haute-Garonne
  - CHU de Montpellier- Hôpital Gui De Chauliac, Montpellier, Hérault
  - CHRU de Tours - Hôpital Bretonneau, Tours, Indre-et-Loire
  - CHRU Nancy, Nancy, Meurthe-et-Moselle
  - CHU de Lille - Hopital Claude Huriez, Lille, Nord
  - Hospices Civils de Lyon - 59 Bd Pinel, Lyon, Rhône
  - Hôpital Pontchaillou, Rennes
- Germany (16):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Epilepsiezentrum Kork, Kehl, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - LMU Klinikum der Universität München - Campus Großhadern, München, Bavaria
  - Epilepsieklinik Tabor, Bernau bei Berlin, Brandenburg
  - Universitätsklinikum Gießen und Marburg GmbH - Standort Marburg, Marburg, Hesse
  - Klinikum Osnabrück GmbH, Osnabrück, Lower Saxony
  - Krankenhaus Mara gGmbH, Bielefeld, North Rhine-Westphalia
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Münster, Münster, North Rhine-Westphalia
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - Kleinwachau Sächsisches Epilepsiezentrum Radeberg Gemeinnützige Gmbh, Radeberg, Saxony
  - Vivantes - Humboldt Klinikum, Berlin
  - Universitätsklinikum Frankfurt, Frankfurt
  - Epilepsie-Zentrum Bodensee, Ravensburg
- Greece (5):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - University General Hospital ''ATTIKON'', Chaïdári
  - University General Hospital of Ioannina, Ioannina
  - AHEPA University General Hospital of Thessaloniki, Thessaloniki
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hungary (4):
  - Pécsi Tudományegyetem Klinikai Kozpont -Ret u., Pécs, Baranya
  - Debreceni Egyetem Klinikai Kozpont Kenezy Gyula Campus, Debrecen, Hajdú-Bihar
  - Budapesti Bajcsy-Zsilinszky Korhaz es Rendelointezet, Budapest
  - SE INK Juhasz Pal Epilepszia Központ, Budapest
- India (5):
  - Nizam's Insti. of Medical Sciences, Hyderabad
  - Mallikatta Neuro Centre, Mangalore
  - Jaslok Hospital and Research, Mumbai
  - Dr G M Taori Memorial CIIMS, Nagpur
  - All India Institute of Medical Sciences (AIIMS), New Delhi
- Italy (17):
  - Università degli Studi G. D'Annunzio Chieti-Pescara, Chieti, Abruzzo
  - Azienda Ospedaliera Universitaria Renato Dulbecco - AO Mater Domini, Catanzaro, Calabria
  - AORN Antonio Cardarelli, Napoli, Campania
  - AUSL di Bologna - Ospedale Bellaria, Bologna, Emilia-Romagna
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genoa, Liguria
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, Lombardy
  - ASST Santi Paolo e Carlo - Azienda Universitaria-Polo Universitario San Paolo, Milan, Lombardy
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino IRCCS, Pavia, Lombardy
  - Azienda Ospedaliero-Universitaria di Modena - Ospedale Civile di Baggiovara, Baggiovara, Modena
  - IRCCS Istituto Neurologico Mediterraneo Neuromed, Pozzilli, Molise
  - Università Politecnica delle Marche Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona, Ancona, The Marches
  - Azienda Ospedaliero Universitaria A Meyer - INCIPIT - PIN, Calambrone, Tuscany
  - Fondazione Policlinico Universitario A Gemelli-Rome, Roma
  - IRCCS Ospedale Pediatrico Bambino Gesù - INCIPIT - PIN, Rome
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona
- Mexico (7):
  - Unidad de Investigación en Salud de Chihuahua S.C.-Mexico city, Mexico City
  - Clinstile, S.A. de C.V., Mexico City
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey
  - Axis Heilsa S. de R.L. de C.V., Obispado
  - Neurociencias Estudios Clinicos S.C., Sinaloa
  - Clinical Research Institute SC-Mexico, Tlalnepantla
  - FAICIC S De RL De CV, Veracruz
- Netherlands (3):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Stichting Epilepsie Instellingen Nederland - Heemstede, Heemstede, North Holland
  - Stichting Epilepsie Instellingen Nederland - Dokter Denekampweg 20, Zwolle, Overijssel
- Poland (15):
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Poznaniu, Poznan, Greater Poland Voivodeship
  - Przychodnia VISTAMED, Wroclaw, Lower Silesian Voivodeship
  - Clinical Best Solutions - Lublin, Lublin, Lublin Voivodeship
  - NZOZ IGNIS dr med. Alicja Lobinska, Świdnik, Lublin Voivodeship
  - Twoja Przychodnia Nowosolskie Centrum Medyczne sp. z o.o, Nowa Sól, Lubusz Voivodeship
  - Santa Familia PTG Lodz, Lodz, Lódzkie
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Neurosphera SP. Z O.O, Warsaw, Masovian Voivodeship
  - Instytut Psychiatrii i Neurologii, Warsaw, Masovian Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - Copernicus Podmiot Leczniczy Sp. z o.o. - ul. Nowe Ogrody 1-6, Gdansk
  - Novo-Med Zielinski i wsp. Sp.J. - ul. Brynowska 44, Katowice
  - Pratia MCM Kraków, Krakow
  - LANDA Specjalistyczne Gabinety Lekarskie, Krakow
  - Premium Clinic Wrocław, Wroclaw
- Portugal (6):
  - ULS de Entre Douro e Vouga, EPE - Hospital de São Sebastião, Santa Maria da Feira, Aveiro District
  - ULS de Matosinhos, EPE - Hospital Pedro Hispano, Senhora da Hora, Porto District
  - Centro Clínico Académico, Braga - Hospital de Braga, Braga
  - ULS de Coimbra, EPE - Hospitais da Universidade de Coimbra, Coimbra
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon
  - Hospital da Luz Torres de Lisboa, Lisbon
- Romania (2):
  - Targu-Mures Emergency Clinical County Hospital - Str. Gh. Marinescu nr.50, Târgu Mureş, Mureș County
  - Emergency University Hospital, Bucharest
- Slovakia (2):
  - IN MEDIC, s.r.o., Bardejov
  - Kraskova 2636, Neurologické oddelenie, Rimavská Sobota
- University Clinical Centre Maribor, Maribor, Slovenia
- South Africa (2):
  - InnoMed Clinical Trial Centre, Cape Town, Western Cape
  - Groote Schuur Hospital, Cape Town, Western Cape
- Spain (18):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Navarra, Pamplona, Navarre
  - CHUVI - H.U. Alvaro Cunqueiro, Vigo, Pontevedra
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Fundacio Assistencial Mutua de Terrassa, Barcelona
  - Hospital Universitario Clínico San Cecilio, Granada
  - Hospital Vithas Granada, Granada
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Ruber Internacional (Grupo Quironsalud), Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Blua Sanitas Valdebebas Hospital, Madrid
  - Hospital blua sanitas valdebebas, Madrid
  - Hospital Regional Universitario de Malaga - Hospital General, Málaga
  - Centro de Neurologia Avanzada, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Klinik Lengg AG, Zurich, Zürich (de), Switzerland
- United Kingdom (8):
  - Morriston Hospital, Swansea, Glamorgan
  - Queen Elizabeth University Hospital-PPDS, Glasgow, Glasgow City
  - Salford Royal Hospital - PPDS, Salford, Manchester
  - The Walton Centre - PPDS, Liverpool, Merseyside
  - University College Hospital, London, Middlesex
  - John Radcliffe Hospital, Oxford, Oxfordshire
  - University Hospital of Wales, Cardiff, South Glamorgan
  - Royal Victoria Infirmary, Newcastle upon Tyne